CLINICAL TRIAL: NCT07372053
Title: Evaluation of an Online Application for Point of Care Ultrasound Training in General Internal Medicine Residents
Status: Not yet recruiting | Type: Observational
Sponsor: Kantonsspital Baden (Other)
Collaborators: Spital Limmattal Schlieren (Other)
Responsible Party: Principal Investigator, Tudor Cosma, Principal Investigator, Kantonsspital Baden
Other Study IDs: 2024-01470
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Point of Care Ultrasound (POCUS); Ultrasound Exam in Emergency/Medical Care; Ultrasound Evaluation
Keywords: POCUS; Point of Care Ultrasound; Point of Care Ultrasonography; Medical Education; Ultrasound Education; POCUS Training; POCUS Education; Ultrasound Supervision; POCUS Supervision; Ultrasound Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POCUS supervision using application: This group is supervised using the online application.
- Usual POCUS supervision: This group receives usual POCUS supervision, without using the application.

SUMMARY:
This study compares Point of Care Ultrasound (POCUS) training in two hospitals, one that uses an online application for supervision and one that does not use the application. The goal of this trial is to learn if POCUS supervision using the online application is associated with improved POCUS skills in residents in General Internal Medicine (GIM). The main question it aims to answer is:

- Do POCUS skills improve more during 6 months in GIM residents supervised using the application than in GIM residents who do not use the application?

Further questions the study aims to answer are:

* Do residents using the application perform more POCUS exams during 6 months than residents not using the application?
* Are residents using the application more satisfied with their POCUS training than residents not using the application?

ELIGIBILITY:
Inclusion Criteria:

* General Internal Medicine resident employed at one of the study sites for at least 2 months
* Probably or definitely interested in achieving POCUS certification (mandatory for the General Internal Medicine specialisation in Switzerland)
* Basic ultrasound course completed (Basic course Abdominal ultrasound or Emergency ultrasound)
* Will spend at least 3 months within a rotation where POCUS training is offered during the 6 months after baseline assessment

Exclusion Criteria:

* Definitely or probably not interested in achieving POCUS certification
* Has already performed more than 80 supervised and more than 160 total POCUS exams
* Will end employment at the study site less than 7 months after baseline assessment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General internal medicine residents at two hospitals in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in POCUS skills | Post-test 6 months (+/- 2 weeks) from pre-test
  POCUS skills will be evaluated on healthy volunteers by video-recorded OSCE

SECONDARY OUTCOMES:
Number of POCUS exams performed | During 6 months after baseline assessment (pre-test)
  In the cohort using the application, the number is automatically recorded. The usual supervision cohort will manually record the number of exams.
Number of supervised POCUS exams performed | During 6 months after baseline assessment (pre-test)
  In the cohort using the application, the number is automatically recorded. The usual supervision cohort will manually record the number of exams.
Number of directly supervised POCUS exams performed | During 6 months after baseline assessment (pre-test)
  Direct supervision means that the supervisor is present during the exam. In the cohort using the application, the number is automatically recorded. The usual supervision cohort will manually record the number of exams.
Change in satisfaction and engagement with POCUS training | Follow-up assessment 6 months (+/- 2 weeks) after baseline assessment
  Measured with a survey
Change in self-assessed POCUS competency | Follow-up assessment 6 months (+/- 2 weeks) after baseline assessment
  Assessed with a survey. Included since the objective evaluation (primary outcome) will not assess all regions that residents are trained to examine, in order to keep the evaluation feasible.

OTHER OUTCOMES:
Usefulness of the online application | 6 months (+/- 2 weeks) after baseline assessment
  Assessed with a survey, only in the cohort using the application
Change from baseline in POCUS skills within the individual cohorts | Post-test 6 month (+/- 2 weeks) from pre-test
  Evaluating how POCUS skills evolve during 6 months in each of the individual study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Wertli, MD PhD, Study Chair — Kantonsspital Baden
Locations (2):
- Switzerland (2):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Spital Limmattal Schlieren, Schlieren, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in compliance with the national and international privacy regulations and after appropriate approval.